CLINICAL TRIAL: NCT04304716
Title: Regional Anesthesia for the Management of Perioperative Pain for Free Flap Reconstruction of the Head and Neck: A Randomized Prospective Trial
Brief Title: Regional Anesthesia for Head and Neck Reconstruction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn from the IRB
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201903261
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Fibular free flap-Block performed (Active Comparator): For subjects in the experimental/regional anesthesia group for anterolateral thigh or radial forearm free flap, during the procedure a catheter will be placed into the donor site (leg or arm), wound bed
  Interventions: Drug: Regional Anesthesia
- Anterolateral thigh free flap-Block performed (Active Comparator): Description: For subjects in the experimental/regional anesthesia group for anterolateral thigh or radial forearm free flap, during the procedure a catheter will be placed into the donor site (leg or arm), wound bed
  Interventions: Drug: Regional Anesthesia
- Radial forearm free flap-Block performed (Active Comparator): Description: For subjects in the experimental/regional anesthesia group for anterolateral thigh or radial forearm free flap, during the procedure a catheter will be placed into the donor site (leg or arm), wound bed
  Interventions: Drug: Regional Anesthesia
- Fibular free flap -Control (No Intervention): No additional procedures beyond the normal standard of care will be performed
- Anterolateral thigh free flap-Control (No Intervention): No additional procedures beyond the normal standard of care will be performed
- Radial forearm free flap-Control (No Intervention): No additional procedures beyond the normal standard of care will be performed

INTERVENTIONS:
Drug: Regional Anesthesia — Block performed is an indwelling wound bed or popliteal catheter placed intraoperatively
  Arms: Anterolateral thigh free flap-Block performed; Fibular free flap-Block performed; Radial forearm free flap-Block performed

SUMMARY:
By utilizing regional anesthesia blocks at the surgery tissue donor sites, it can potentially reduce post-operative pain while also reducing the use of opioids. It can aim to measure the reduction in opioid use, reduction in pain scores, patient satisfaction, and because there is not a current protocol established for regional anesthesia use for free flap reconstruction, and we aim to standardize the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing microvascular fibula free flap reconstruction of the head and neck
* Subjects undergoing primary reconstruction for both benign and malignant etiology

Exclusion Criteria:

* Pregnant women
* Subjects with true allergies to the study drugs, reporting anaphylaxis in the past
* Subjects undergoing reconstruction with more than 1 free flap
* Subjects undergoing secondary reconstructions
* Subjects undergoing surgery for osteonecrosis
* History of enrollment in a pain management program
* Any subject currently enrolled in pain management, or currently taking long acting opioids such as methadone or oxycontin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 72 hours (3 days) post-operatively
  Subjects' morphine equivalent dose. Postoperative period commences at extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Fernandes, MD, DMD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States